CLINICAL TRIAL: NCT00464165
Title: Comparison of the Efficacy and Safety of 2 Oral Doses of Rimonabant, 5mg/Day or 20mg/Day, Versus Placebo, as an Aid to Smoking Cessation; Multiple Country, Randomized, Double-blind, 3-arm, 10-week Treatment, 40-week Follow-up
Brief Title: Comparison of Efficacy and Safety of Rimonabant 5mg/Day or 20mg/Day Versus Placebo in Smoking Cessation
Acronym: STRATUS-EU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4474; SR141716
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Smoking Cessation
Keywords: abstinence
MeSH Terms: conditions — Smoking Cessation | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant

SUMMARY:
The primary objective is to assess the efficacy of 2 fixed doses of rimonabant versus placebo on abstinence from tobacco use in cigarette smokers.

The secondary objective is to evaluate the effects of rimonabant on craving and weight and on the clinical and biological safety and tolerability of rimonabant in a population of cigarette tobacco smokers during a 10-week treatment period and to observe the percentage of abstinent subjects during a 40-week follow-up post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Smokers smoking at least 10 cigarettes/day as a mean within the 2 months preceding the screening visit
* Motivated to quit with a score greater than or equal to 6 on the ten-point Motivation Scale

Exclusion Criteria:

* Non tobacco cigarettes consumption
* Chronic use of marijuana
* Pregnancy, breastfeeding
* Any clinically significant disease that might interfere with the efficacy or safety evaluation of the study drug
* Concomitant use of drugs as an aid to smoking cessation or that might induce weight change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2002-11; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence from smoking during the last 4 weeks of treatment reported by the subject and confirmed by exhaled carbon monoxide (CO) and cotinine measurements

SECONDARY OUTCOMES:
Efficacy: mean change of the total score of Questionnaire on Smoking Urges (QSU) brief scale, categorical change in body weight in subjects with Body Mass Index lower than 30 kg/m² at baseline who achieve prolonged abstinence
Safety data

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom